CLINICAL TRIAL: NCT02970825
Title: Move and Feel Good : Effects of Intensive Physical Training on Brain Plasticity, Cognition and Psychological Well-being. "Effets de l'entraînement Physique Intensif Sur la plasticité cérébrale, la Cognition et le Bien être Psychologique".
Brief Title: Move and Feel Good : Effects of Intensive Physical Training on Brain Plasticity, Cognition and Psychological Well-being.
Acronym: Move&FG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Anne G. De Volder, MD, PhD, MD, PhD, Senior Research Associate, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Etude 2016/17FEV/060
Record Dates: First submitted 2016-10-09; First posted 2016-11-22 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Learning Disorders; Depression; Anxiety
Keywords: exercise medicine; youth; adolescents; students
MeSH Terms: conditions — Learning Disabilities; Depression; Anxiety Disorders | interventions — Exercise; Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: Two experimental arms: physical training and relaxation program, including social activities. Both programs are conducted in parallel with adolescents and young people.
  A first study was conducted among schoolchildren and was published. The second study was conducted in a clinical population of Area + -Fond'Roy psychiatric hospital in Brussels. Both studies were performed in a parallel order and randomized at the beginning of the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): The experimental, intensive exercise regime will include 50-min sessions four times a week during five weeks (for a total of about 17 hours) combining structured aerobic exercise (at least 20 minutes jogging and moderate to high intensity active games) and anaerobic lactic resistance exercise (power training with gymn weights).
  Interventions: Other: Exercise
- Relaxation (Active Comparator): The control activity will include 50-min sessions four times a week during five weeks (for a total of about 17 hours) combining mindfulness, stretching and low intensity active games (breath control, proprioception, walking, social relaxation, flexibility training).
  Interventions: Other: Relaxation

INTERVENTIONS:
Other: Exercise — Moderate to high intensity physical training
  Other Names: Physical training
  Arms: Exercise
Other: Relaxation — Low intensity physical activity and relaxation
  Other Names: Flexibility training
  Arms: Relaxation

SUMMARY:
The investigators perform a prospective, randomized, clinical study involving students in education with mood disorders and randomized to an intensive exercise program or a control relaxation activity.

DETAILED DESCRIPTION:
The investigators wish to document the benefit of an intensive and structured exercise program in youth with the aim to identify the most effective programs that can improve psychological well-being, especially reducing depressive and anxiety symptoms and improving self-esteem. This study targets participants aged 9 to 30 years and included in an education program (from 4th Grade to undergraduate university or college). The investigators propose to perform a prospective, randomized, clinical study involving participants with mood disorders (International Classification of Diseases, 10th Revision, Clinical Modification (ICD-10-CM) for medical coding: ICD-10-CM F32.9), anxiety (ICD-10-CM F41.9), specific learning disabilities (ADHD hyperactivity (ICD-10-CM F90.2), dyslexia-dyscalculia-dyspraxia (ICD-10-CM F81.0, F81.2, F81.81)) and healthy subjects equally distributed for confounding variables (age, gender, subclinical or clinical depressive symptoms). The participants (ambulatory or inpatients) will be enrolled either in an experimental, intensive and structured aerobic exercise regime or in a active control activity of stretching and relaxation conducted in parallel. The effects of this program will be assessed for i) psychological symptoms, using questionnaires, ii) cognitive function, particularly attention skills and executive functions, in neuropsychological tasks, and iii) physical abilities (through physical testing). To investigate the therapeutic value of exercise in the prevention of depressive and anxiety symptoms and in the treatment of mood disorders in the young student is a necessity imposed by the current outbreak of depression among adolescents and young people at school. To promote the exercise medicine based on the level of evidence in this specific domain, rigorous experimental studies must be performed. Depending on the results, a medical imaging will be proposed to participants at the end of the behavioral study. This will be a functional magnetic resonance imaging in physiological activation condition (performing a behavioral task such as a Stroop task suited to the subject's age), performed before and after intensive physical training.

ELIGIBILITY:
Inclusion Criteria:

* involved in education program
* absence of contra-indication of physical activity
* does accept randomization
* no history of neurological illness or brain trauma
* no history of psychiatric illness (exclusion of psychotic symptoms)
* absence of contra-indication to magnetic resonance imaging
* no uncorrected sensory impairment (must understand the therapist)
* absence of conduct disorders (violence, school bullying)

Exclusion Criteria:

* does not provide informed consent
* unstable diabetes
* Body mass index above P95 (or above 30 for adults) (except medical authorization)
* coagulation disorders
* severe and unstable asthma
* history of hearth malformation or heart disease
* medical conditions prohibiting sport or contraindicating physical activity

Ages: 9 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2021-11-18 (Estimated); Study Completion 2021-11-18 (Estimated)

PRIMARY OUTCOMES:
Change from baseline psychological well-being as assessed using depression and anxiety questionnaires | at 3 weeks, at 6 weeks and through study completion, up to 6 months
  Hospital Anxiety Depression Scale (HADS) in french version for all participants, mainly suitable for inpatients
Change from baseline psychological well-being as assessed using self-esteem, mood and anxiety questionnaires | at 3 weeks, at 6 weeks and through study completion, up to 6 months
  State-Trait Anxiety Inventory (STAI) in french version for all participants, mainly suitable for outpatients

SECONDARY OUTCOMES:
Change from baseline psychological well-being as assessed using depression questionnaires for children | at 3 weeks, at 6 weeks and through study completion, up to 6 months
  Children's Depression Inventory (CDI) in french version
Change from baseline psychological well-being as assessed using depression questionnaires for adolescents and adults | at 3 weeks, at 6 weeks and through study completion, up to 6 months
  Beck Depression Inventory (BDI-13) in french version
Change from baseline psychological well-being as assessed using depression questionnaire for young people and adults | at 3 weeks, at 6 weeks and through study completion, up to 6 months
  Self-depression scale (SDS) in french version
Change from baseline psychological well-being as assessed using self-esteem questionnaires | at 3 weeks, at 6 weeks and through study completion, up to 6 months
  Self-perception profile for children or adolescents in french version
Change from baseline physical condition : size | at 3 weeks, at 6 weeks and through study completion, up to 6 months
  Height in meters
Change from baseline physical condition : weight | at 3 weeks, at 6 weeks and through study completion, up to 6 months
  Weight in kilograms
Change from baseline physical condition as assessed in bioelectrical impedance analysis | at 3 weeks, at 6 weeks and through study completion, up to 6 months
  Body mass index (BMI) in kilograms divided by the square of the height in meters (kg/m2)
Change from baseline physical condition : body muscle ratio | at 3 weeks, at 6 weeks and through study completion, up to 6 months
  Body muscle percentage : {body muscle mass (kg) / total body mass (kg)} x 100
Change from baseline physical condition : body fat ratio | at 3 weeks, at 6 weeks and through study completion, up to 6 months
  Body fat percentage : {body fat mass (kg) / total body mass (kg)} x 100
Change from baseline physical condition as assessed using field running tests or a cycle ergometer | at 3 weeks, at 6 weeks and through study completion, up to 6 months
  An estimation of maximal oxygen consumption in field running test (20m-beep test).
  A submaximal effort test using a cycle ergometer.
Change from baseline cognitive function as assessed using computerized neuropsychological testing of cognitive control | at 3 weeks, at 6 weeks and through study completion, up to 6 months
  Attention and conflict resolution testing using a variant of the Eriksen Flanker task, adapted for age, in E-Prime.
Change from baseline cognitive function as assessed using computerized neuropsychological testing of inhibitory control | at 3 weeks, at 6 weeks and through study completion, up to 6 months
  Inhibitory control testing using a go-no go test adapted in E-Prime.

CONTACTS AND LOCATIONS:
Overall Officials: Anne G De Volder, MD, PhD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Université catholique de Louvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
This is a monocentric study. All individual participant data that allow subject identification will be kept confidential.

REFERENCES:
- [Derived] Philippot A, Meerschaut A, Danneaux L, Smal G, Bleyenheuft Y, De Volder AG. Impact of Physical Exercise on Symptoms of Depression and Anxiety in Pre-adolescents: A Pilot Randomized Trial. Front Psychol. 2019 Aug 8;10:1820. doi: 10.3389/fpsyg.2019.01820. eCollection 2019. PMID 31440186